CLINICAL TRIAL: NCT03116659
Title: CTCL Directed Therapy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ali Dana, Dermatologist, James J. Peters Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAN-15-028
Record Dates: First submitted 2017-04-11; First posted 2017-04-17 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Lymphoma, T-Cell, Cutaneous
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — Doxycycline; Imiquimod

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm (Experimental): Doxycycline 100 mg PO BID x 14 days, then Imiquimod up to 2 packs 3/ week x 28 days
  Interventions: Drug: Doxycycline; Drug: Imiquimod

INTERVENTIONS:
Drug: Doxycycline — Doxycycline 100 mg PO BID x 14 days
Drug: Imiquimod — up to 2 packs 3/ week x 28 days

SUMMARY:
Cutaneous lymphomas are rare cancers of lymphocytes (white blood cells) that involve the skin. Mycosis Fungoides (MF) is the most common type of Cutaneous T-cell lymphoma (CTCL) that typically presents with red, scaly patches that often mimic eczema or chronic dermatitis. The incidence of MF is about 1/100,000. Skin lesions tend to appear before the diagnosis of CTCL is made by several years. Early skin lesions may look like any dermatitis, eczema, or psoriasis, leading to delays in the diagnosis.

Inflammation secondary to bacterial infection is thought to contribute to the T-cell proliferation in this type of cutaneous T-cell lymphoma. Antibiotic use for other purposes has shown to reduce the inflammation and size of lesions in CTCL patients. There has been limited studies with the use of antibiotics as direct treatment for this cancer.

Host immunity is important in decreasing cancer development and progression. Imiquimod is a molecule that stimulates host immunity to reduce the progression of CTCL. There is strong evidence of clinical efficacy such that the National Comprehensive Cancer Network (NCCN) guidelines recommend Imiquimod for CTCL. Imiquimod is available in generic form, making it unlikely to be registered specifically for CTCL, despite its efficacy.

Additionally, imiquimod is considered a first line treatment according to National Comprehensive Cancer Network (NCCN) guidelines for the treatment of Mycosis Fungoides.

There are currently no studies that have been published that address treating CTCL patients with a combined approach of 1) decreasing inflammation caused by bacterial with antibiotics, and 2) enhancing the host immune system to destroy cancer cells. Our theory is if we treat patient with 14days of antibiotics and 30 days of Imiquimod there will be significant reduction in skin lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 30 - 89 years old
* Stages I to II CTCL patients
* Normal renal function, Cr ≤ 1.5

Exclusion Criteria:

* Aggressively progressing CTCL
* Active infection and/or concurrent malignancy
* Poor renal function (Cr > 1.5)
* Pregnancy (HCG serum +)
* History of bone marrow suppression, MDS, anemia (Hemoglobin < 8), thrombocytopenia (< 50,000) or neutropenia (ANC < 1500)
* CHF, MI within last 6 months
* Endocarditis
* Allergies to Imiquimod or doxycycline

Ages: 30 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Pilot assessment of response. | 1 year
  Pilot assessment of response assessed by decreased size or surface change of the 5 lesions

CONTACTS AND LOCATIONS:
Overall Officials: Ali Dana, MD, Principal Investigator — James J. Peters VAMC
Locations (1):
- James J Peters Bronx Veterans Affairs Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Del Guzzo CA, Kojadinovic A, Vinnakota RR, Geskin LJ, Newman JC, Langhoff E, Park YA, Bates SE, Dana AN. Antibiotics and Imiquimod for Cutaneous T-Cell Lymphoma in Veterans: A Patient Population with Agent Orange Exposure. Oncologist. 2021 Sep;26(9):727-e1488. doi: 10.1002/onco.13785. Epub 2021 May 14. PMID 33851477